CLINICAL TRIAL: NCT01829607
Title: Functional Electrical Stimulation of Peripheral Muscles in Heart Failure With Preserved Left Ventricular Ejection Fraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, John Parissis, Assistant Professor of Cardiology, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FES-HFPEF
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Heart Failure With Preserved Left Ventricular Ejection Fraction

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Functional electrical stimulation (Active Comparator): Functional electrical stimulation of lower limbs
  Interventions: Other: Functional electrical stimulation of peripheral muscles
- Placebo (Placebo Comparator)

INTERVENTIONS:
Other: Functional electrical stimulation of peripheral muscles
  Arms: Functional electrical stimulation

SUMMARY:
The purpose of this study is to evaluate the effects of functional electrical stimulation of peripheral muscles on clinical and emotional status, endothelial function and left ventricular diastolic function in heart failure with preserved left ventricular ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

(i) symptoms [New York Heart Association (NYHA) class II or III] and signs typical of heart failure

(ii) left ventricular (LV) ejection fraction (LVEF) >50% and LV end-diastolic volume index <97 mL/m2

(iii) findings of left atrial (LA) dilatation (LA volume index >40mL/m2), LV hypertrophy and/or LV diastolic dysfunction [ie, mitral E/A ratio <1 or >2, mitral E/e' ratio >15 or 8-15, (A pulmonary - A mitral) duration difference >30 ms etc)

(iv) no alterations in medical therapy during the previous 4 weeks

(v) no myocardial infarction within 3 months prior to enrollment

Exclusion Criteria:

recent (≤4 weeks) heart failure decompensation

* acute coronary syndrome
* chronic inflammatory diseases and malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | Six weeks
Quality of life | Six weeks
Emotional status | Six weeks

SECONDARY OUTCOMES:
Left ventricular diastolic function | Six weeks
Endothelial function | Six weeks

OTHER OUTCOMES:
Neurohormonal activation | Six weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Attikon University Hospital, Athens, Greece

REFERENCES:
- [Derived] Karavidas A, Driva M, Parissis JT, Farmakis D, Mantzaraki V, Varounis C, Paraskevaidis I, Ikonomidis I, Pirgakis V, Anastasiou-Nana M, Filippatos G. Functional electrical stimulation of peripheral muscles improves endothelial function and clinical and emotional status in heart failure patients with preserved left ventricular ejection fraction. Am Heart J. 2013 Oct;166(4):760-7. doi: 10.1016/j.ahj.2013.06.021. Epub 2013 Aug 30. PMID 24093858